CLINICAL TRIAL: NCT05330546
Title: Evaluation of the Stability of Implants Placed in Low Quality Bone Following the Use of Osseodensification Technique Versus Ridge Expanders: Randomized Clinical Trial
Brief Title: Evaluation of Implant Stability in Low Quality Bone Following the Use of Osseodensifiers Versus Ridge Expanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Samir Nabih, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12722
Record Dates: First submitted 2022-04-02; First posted 2022-04-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2022-09

CONDITIONS: Low Bone Density
Keywords: osseodensification; ridge expansion screw
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osseodensification technique group (Experimental): 10 patients will be randomly assigned to the osseodensification group so the implant osteotomy will be prepared using densah burs
  Interventions: Procedure: Densah burs
- Ridge expansion screw group (Active Comparator): 10 patients will be randomly assigned to the ridge expansion screw group so the implant osteotomy will be prepared using ridge expansion screws
  Interventions: Procedure: Ridge expansion screws

INTERVENTIONS:
Procedure: Densah burs — using Densah burs to prepare implant osteotomy
  Arms: Osseodensification technique group
Procedure: Ridge expansion screws — using Ridge expansion screws to prepare implant osteotomy
  Arms: Ridge expansion screw group

SUMMARY:
the use of osseodensification technique compared to ridge expansion screws in low bone quality

DETAILED DESCRIPTION:
using Densah burs in preparation of implant osteotomy compared to ridge expansion screws in low quality bone

ELIGIBILITY:
Inclusion Criteria:

* • Single tooth missing in the maxillary region with D3 (350-850 HU) and D4 (150-350 HU) bone (Sultana et al., 2020).

  * A minimum of 4 mm residual buccolingual bone width at site of implant placement (Koutouzis et al., 2019).

    * The recipient site of the implant should be free from any pathological conditions.
    * No diagnosed bone disease or medication known to affect bone metabolism.
    * Patients who are cooperative, motivated and hygiene conscious.
    * Patients having adequate inter-occlusal space of 8-10 mm (Fernández et al., 2017)

Exclusion Criteria:

* Systemic conditions/diseases that contraindicate surgery (Jarikian et al., 2021).

  * Patients who have any habits that might jeopardize the osseointegration process, such as current smokers (Vollmer et al., 2020).
  * Patients with parafunctional habits that produce overload on implant, such as bruxism and clenching (Sultana et al., 2020).
  * Alcohol or drug abuse (Ibrahim et al., 2020).
  * Pregnant and lactating women.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Implant stability | change from baseline at 3 month
  assessing the stability using Osstell
Implant stability | change from baseline at 6 month
  assessing the stability using Osstell

SECONDARY OUTCOMES:
Radiographic bone density | change from baseline at 3 month
  using CBCT in mm
Radiographic bone density | change from baseline at 6 month
  using CBCT in mm
Change in crestal bone level | change from baseline at 3 month
  using CBCT in mm
Change in crestal bone level | change from baseline at 6 month
  using CBCT in mm
Change in buccolingual bone width | change from baseline at 3 month
  using CBCT in mm
Change in buccolingual bone width | change from baseline at 6 month
  using CBCT in mm
Patient reported outcomes | at time of surgery
  10 mm Visual analogue scale from 1 to 10 with 1 minimal pain and 10 worst pain experience

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Barbary, Assis. prof., Principal Investigator — Main supervisor
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
raw data will be shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: upon request for 2 days
Access Criteria: file including the raw data

REFERENCES:
- [Derived] Nabih MS, Ashour OAM, Abbas WM, ElBarbary A. Evaluation of the stability of implants placed in low-quality bone following the use of osseodensification technique versus ridge expanders:randomized clinical trial. BMC Oral Health. 2025 Sep 17;25(1):1413. doi: 10.1186/s12903-025-06918-y. PMID 40963121